CLINICAL TRIAL: NCT04699435
Title: Effect of the Duration of Pre-oxygenation (3 Minutes vs 6 Minutes) on Apnea Tolerance in Obese Patients (BMI> 30 kg / m2) During the Induction of General Anesthesia
Brief Title: Effect of the Duration of Pre-oxygenation on Apnea Tolerance in Obese Patients During the Induction of General Anesthesia
Acronym: OBE_PreOx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OBE_PreOx
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Patients with a BMI <25 kg / m² requiring general anesthesia with a pre-oxygenation for 3 minutes
  Interventions: Other: Control
- PreOx_3min (Experimental): Patients with a BMI between 30 kg / m² and 40 kg / m² requiring general anesthesia randomized to the pre-oxygenation group for 3 minutes
  Interventions: Other: PreOx_3min
- PreOx_6min (Experimental): Patients with a BMI between 30 kg / m² and 40 kg / m² requiring general anesthesia randomized to the pre-oxygenation group for 6 minutes
  Interventions: Other: PreOx_6min

INTERVENTIONS:
Other: Control — All patients are installed with a 30 ° proclive and have pre-oxygenation (FiO2 = 1) with a face mask. At the end of the 3-minute pre-oxygenation for the "Control" group, the values of ORI, SpO2, mean arterial pressure and heart rate are recorded.
  Arms: Control
Other: PreOx_3min — Patients with a BMI between 30 kg / m² and 40 kg / m² are distributed according to a random allocation in the group "PreOx_3min".
  All patients are installed with a 30 ° proclive and have pre-oxygenation (FiO2 = 1) with a face mask. At the end of the 3-minute pre-oxygenation for the "PreOx_3min" group, the values of ORI, SpO2, mean arterial pressure and heart rate are recorded.
  Arms: PreOx_3min
Other: PreOx_6min — Patients with a BMI between 30 kg / m² and 40 kg / m² are distributed according to a random allocation in the group "PreOx_6min".
  All patients are installed with a 30 ° proclive and have pre-oxygenation (FiO2 = 1) with a face mask. At the end of the 6-minute pre-oxygenation for the "PreOx_3min" group, the values of ORI, SpO2, mean arterial pressure and heart rate are recorded.
  Arms: PreOx_6min

SUMMARY:
The occurrence of arterial oxygen desaturation (hypoxemia) during the induction of general anesthesia remains one of the main causes of complications and mortality in anesthesia. In a healthy patient breathing in ambient air [Inspired O2 fraction (FiO2) = 21%] before the onset of narcosis, a drop in arterial O2 saturation (SpO2) occurs within 1 to 2 minutes. When pre-oxygenation is performed for 3 minutes in healthy subjects with FiO2 = 100%, SpO2 is less than 97% after 7.9 minutes of apnea and arterial O2 desaturation (SpO2 <93%) occurs after 8 to 9 minutes. For this reason and "in order to prevent arterial desaturation during tracheal intubation or supraglottic device insertion maneuvers", it is recommended "to systematically perform a pre-oxygenation procedure (3 min / 8 deep breaths) , including in the context of an emergency ". Tolerance to apnea is conditioned by the amount of O2 stored during the pre-oxygenation phase. Oxygen is transported to different tissues in 2 forms: combined with hemoglobin (Hb) and in dissolved form. In ambient air, the quantity of O2 transported by the Hb is much greater than the part transported in dissolved form. However, when the patient breathes a gas enriched in O2, all the molecules of Hb are quickly saturated (SpO2 = 100%), while the content of dissolved O2 increases constituting a reserve allowing to increase the tolerance to apnea.

Under usual conditions (3 minutes pre-oxygenation with FiO2 = 1), tolerance to apnea is shorter in obese subjects. Arterial O2 desaturation occurs after 2-3 minutes of apnea in patients with grade III obesity [Body Mass Index (BMI)> 35 kg / m2]. In addition, arterial O2 desaturation is faster the higher the BMI is. In fact, in obese patients, the lung volumes that can be mobilized in the supine position are modified compared to the non-obese subject: decrease in vital capacity, decrease in expiratory reserve volume, increase in airway resistance, decrease in thoracic compliance. These changes are, in part, explained by the weight of tissue on the rib cage and abdomen leading to compression of the lungs and diaphragm. In addition, there is also an increase in oxygen consumption in patients with a BMI> 40.

Different techniques have been proposed to increase apnea tolerance in obese patients. For Dixon et al., The desaturation of the morbidly obese subject (BMI> 40 kg / m2) is less rapid after 3 minutes of pre-oxygenation carried out with the patient in a half-seated position at 25 °: 201 seconds against 155 seconds in the Control group. This additional time seems to correlate with the value of the arterial pressure in O2 (PaO2) measured at the end of the pre-oxygenation (442 vs 360 mmHg). Likewise, the proclive position (30 ° reverse Trendelenburg) during the pre-oxygenation phase seems effective in limiting the occurrence of desaturation after induction.

The O2 reserve is usually assessed by measuring the partial pressure of O2 in the arterial blood. A value greater than 100 mmHg indicates that an amount of O2 is "in reserve", increasing tolerance to apnea. In practice, this examination is not feasible in current practice because it requires the performance of an invasive procedure, cannot be measured continuously and the rendering of the result is delayed by several minutes. In recent years, a technology based on spectrophotometry has been developed to measure the saturation of Hb in O2 in non-pulsatile blood. By algorithmic transformation, an Oxygen Reserve Index (ORI) is calculated. Its value varies from 0 to 1 and covers a data range between 100 and 200 mmHg of blood pressure in O2 (moderate hyperoxia). This data is obtained continuously and non-invasively from a sensor (RD Rainbow SET R Sensors; Masimo) placed on the 3rd or 4th finger of the hand. When a patient receives an O2 enriched gas mixture, the value of ORI increases rapidly and reaches a plateau. When the patient is in apnea, the drop in the ORI value precedes the drop in SpO2 by several tens of seconds. In a pilot study observing the kinetics of ORI in non-obese (BMI <25 kg / m2) or obese (BMI> 30 kg / m2) anesthetized patients, we observed that the time required to reach the plateau of l The ORI was longer (133 ± 30 seconds) in "obese" patients compared to "non-obese" patients (89 ± 28 seconds). Thus, one hypothesis to explain the poorer tolerance to apnea in obese patients would be that the duration of 3 minutes of pre-oxygenation as recommended in the recommendations is insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient to have general anesthesia
* Patient affiliated to a health insurance plan
* French-speaking patient
* Patient who has given free, informed and written consent

Exclusion Criteria:

* Patient with a BMI between 25 and 30 kg / m2
* Patient with a BMI> 40 kg / m2
* Patient whose O2 stock is insufficient, without this being linked to obesity
* Patient with severe respiratory pathology (COPD stage 3 or 4, severe asthma)
* Patient with active smoking
* Patient with a history of lobectomy or pneumonectomy
* Patient coming for emergency surgery
* Patient with a known allergy to rocuronium or sufentanil or propofol
* Pregnant or breastfeeding women
* Patient under guardianship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Apnea tolerance | End of pre-oxygenation 3 min versus 6 min
  This outcome is to compare the duration of apnea tolerance (SpO2 value ≤ 94%) in obese patients (30 kg / m2 <BMI <40 kg / m2) depending on the duration of pre-oxygenation (3 minutes vs 6 minutes) during induction of general anesthesia compared to non-obese subjects (BMI <25 kg / m2).

SECONDARY OUTCOMES:
ORI profile | End of pre-oxygenation 3 min versus 6 min
  This outcome is to evaluate ORI profile in obese patients according to the duration of pre-oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ALFONSI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph, France

REFERENCES:
- [Result] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Result] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Result] Gambee AM, Hertzka RE, Fisher DM. Preoxygenation techniques: comparison of three minutes and four breaths. Anesth Analg. 1987 May;66(5):468-70. No abstract available. PMID 3578856
- [Result] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Result] Berthoud MC, Peacock JE, Reilly CS. Effectiveness of preoxygenation in morbidly obese patients. Br J Anaesth. 1991 Oct;67(4):464-6. doi: 10.1093/bja/67.4.464. PMID 1931404
- [Result] Tsymbal E, Ayala S, Singh A, Applegate RL 2nd, Fleming NW. Study of early warning for desaturation provided by Oxygen Reserve Index in obese patients. J Clin Monit Comput. 2021 Aug;35(4):749-756. doi: 10.1007/s10877-020-00531-w. Epub 2020 May 18. PMID 32424516